CLINICAL TRIAL: NCT03120598
Title: Substance Abuse Treatment to HIV Care (SAT2HIV): The Implementation & Sustainment Facilitation Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SAT2HIV-ISF; R01DA038146 (NIH)
Record Dates: First submitted 2017-04-18; First posted 2017-04-19 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Substance Use
Keywords: preparation strategies; implementation strategies; sustainment strategies
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATTC strategy (Active Comparator): Behavioral: Addiction Technology Transfer Center (ATTC) strategy: A staff-focused strategy that includes 10 discrete strategies (e.g., centralized technical assistance, conduct educational meetings, provide ongoing consultation).
  Interventions: Behavioral: ATTC strategy
- ISF strategy (Experimental): Behavioral: Implementation & Sustainment Facilitation (ISF) strategy: An organization-focused strategy that includes 7 discrete strategies (e.g., use of an implementation advisor, organize implementation team meetings, conduct cyclical small tests of change) and Addiction Technology Transfer Center (ATTC) strategy: A staff-focused strategy that includes 10 discrete strategies (e.g., centralized technical assistance, conduct educational meetings, provide ongoing consultation).
  Interventions: Behavioral: ATTC strategy; Behavioral: ISF strategy

INTERVENTIONS:
Behavioral: ATTC strategy — Addiction Technology Transfer Center (ATTC) strategy: A staff-focused strategy that includes 10 discrete strategies (e.g., centralized technical assistance, conduct educational meetings, provide ongoing consultation).
Behavioral: ISF strategy — Implementation & Sustainment Facilitation (ISF) strategy: An organization-focused strategy that includes 7 discrete strategies (e.g., use of an implementation advisor, organize implementation team meetings, conduct cyclical small tests of change).
  Arms: ISF strategy

SUMMARY:
A cluster randomized experiment focused on testing the extent to which the organization-focused Implementation & Sustainment Facilitation (ISF) strategy is an effective adjunct to the staff-focused Addiction Technology Transfer Center (ATTC) strategy.

DETAILED DESCRIPTION:
A cluster randomized experiment with 39 AIDS service organizations located across the United States. The overarching goal is to test the extent to which the organization-focused Implementation & Sustainment Facilitation (ISF) strategy is an effective adjunct to the staff-focused Addiction Technology Transfer Center (ATTC) strategy.

ELIGIBILITY:
Inclusion Criteria:

* AIDS service organizations have to

  1. serve a minimum of 100 individuals living with HIV/AIDS per year,
  2. have at least two frontline staff who were willing and able to be trained in the Motivational Interviewing-based Brief Intervention (MIBI) Experiment's MIBI for substance use, and
  3. have at least one leadership staff (i.e., supervisor, manager, director) willing and able to help ensure case-managers were given sufficient time for project participation.

     Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Time-to-Proficiency (TTP) Score | Assessed at the end of the 2-month post-workshop preparation phase
  A continuous measure representing the number of days between completion of the training workshop by targeted staff and targeted staff's demonstration of proficiency in the motivational interviewing-based brief intervention.
Implementation Effectiveness Index (IEI) Score | Assessed at the end of the 6-month implementation phase
  A continuous measure representing the sum of the standardized cumulative number of motivational interviewing brief interventions delivered by targeted staff (i.e., consistency) and the cumulative integrity score of targeted staff's delivered of the motivational interviewing-based brief intervention (i.e., quality).
Level of Sustainment (LOS) Score | Assessed at the end of the 6-month sustainment phase
  A continuous measure representing the number of Motivational Interviewing-based Brief Interventions targeted Brief Intervention Staff report delivery of the motivational interviewing-based brief intervention during the past 6-months following the end of the implementation phase.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Garner, PhD, Principal Investigator — RTI International
Locations (39):
- United States (39):
  - HIV Care Directions, Phoenix, Arizona
  - Foothill AIDS Project, Claremont, California
  - AIDS Services Foundation, Orange County, Irvine, California
  - AIDS Project Los Angeles, Los Angeles, California
  - Shanti, San Francisco, California
  - AIDS Project Greater Danbury, Inc., Danbury, Connecticut
  - AIDS Connecticut, Inc., Hartford, Connecticut
  - Delaware HIV Consortium, Wilmington, Delaware
  - The Women's Collective, Washington D.C., District of Columbia
  - Project Response, Inc., Melbourne, Florida
  - Live Forward (AIDS Athens), Athens, Georgia
  - Champaign-Urbana Public Health District (CUPHD), Champaign, Illinois
  - The Project of the Quad Cities (TPQC), Davenport, Iowa
  - AIDS Volunteers, Inc. (AVOL), Lexington, Kentucky
  - Southwest Louisiana AIDS Council, Lake Charles, Louisiana
  - AIDS Project Worcester, Worcester, Massachusetts
  - Health Emergency Lifeline Programs (HELP), Detroit, Michigan
  - Community Health Awareness Group (CHAG), Detroit, Michigan
  - Community AIDS Resources and Education Services (CARES), Kalamazoo, Michigan
  - Minnesota AIDS Project, Minneapolis, Minnesota
  - Burrell Behavioral Health, Springfield, Missouri
  - Doorways, St Louis, Missouri
  - Places for People (p4p), St Louis, Missouri
  - Project ARK, St Louis, Missouri
  - St. Louis Effort For AIDS (EFA), St Louis, Missouri
  - Nebraska AIDS Project (NAP), Omaha, Nebraska
  - Southern NH HIV/AIDS Task Force a.k.a. NH Partnership, Nashua, New Hampshire
  - Caracole House, Cincinnati, Ohio
  - ARC Ohio, Columbus, Ohio
  - HIV Alliance, Eugene, Oregon
  - AID Upstate, Greenville, South Carolina
  - Chattanooga CARES, Chattanooga, Tennessee
  - Nashville CARES, Nashville, Tennessee
  - Panhandle AIDS Support Organization, Amarillo, Texas
  - Triangle Area Network, Beaumont, Texas
  - AIDS Foundation Houston, Houston, Texas
  - Alamo Area Resource Center, San Antonio, Texas
  - Utah AIDS Foundation, Salt Lake City, Utah
  - Vermont CARES, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garner BR, Zehner M, Roosa MR, Martino S, Gotham HJ, Ball EL, Stilen P, Speck K, Vandersloot D, Rieckmann TR, Chaple M, Martin EG, Kaiser D, Ford JH 2nd. Testing the implementation and sustainment facilitation (ISF) strategy as an effective adjunct to the Addiction Technology Transfer Center (ATTC) strategy: study protocol for a cluster randomized trial. Addict Sci Clin Pract. 2017 Nov 17;12(1):32. doi: 10.1186/s13722-017-0096-7. PMID 29149909